CLINICAL TRIAL: NCT02854449
Title: Biomarkers of Tumor Response in Hypofractionated Radiotherapy
Brief Title: Tumor Response in Hypofractionated Radiotherapy
Acronym: TRHR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Celia, Doctor, Peking University First Hospital
Other Study IDs: 20161022
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Neoplasms
Keywords: Immune Marker; Immunologic Marker; Radiotherapy; Dose Hypofractionation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will follow-up different immune cell populations in the blood before, during and after high dose radiation therapy which should give new information of the efficacy of Local Hypofractionated Radiotherapy and a rationale for adjuvant immunotherapy.

DETAILED DESCRIPTION:
* Patient information and collection of a signed informed consent form
* Clinical data collection
* Blood samples of 5 mL:

  1. after registration, prior to the first fraction of radiotherapy
  2. during radiotherapy sessions
  3. one month, 3 months after the last radiotherapy session
* Storage of the blood samples at ambient temperature
* Transportation of the samples to the Institute of Biology of Lille (IBL) - CNRS UMR8161 for analysis
* Destruction of the samples at the end of the analysis

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a hypofractionated irradiation;
* pathologically confirmed Unspecified Adult Solid Tumor
* Age ≥ 18 years old
* KPS≥70
* Signed written informed consent.

Exclusion Criteria:

* Patient treated by chemotherapy, targeted or immunotherapy within 21 days before the first sampling,
* Pregnant or breastfeeding woman,
* Patient under guardianship or tutorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receive local hypofractionated radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of immune cells | prior to the first fraction of radiotherapy;14(±2) days from the begining of RT; the day (±2) of the last radiotherapy sessions ;one month, 3 months after the last radiotherapy session
  The primary endpoint is the change of the percentage of immune cells before, during and after radiotherapy

SECONDARY OUTCOMES:
Local control | 3 months
  Local control of radiotherapy will be assessed based on Response Evaluation Criteria in Solid Tumors(RECIST)1.1
Acute and Late toxicities | 3 months
  Acute and late toxicities will be assessed based on the common toxicity criteria for adverse events version 4.0 (CTCAEv4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Gao Xianshu, Master, Study Chair — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No